CLINICAL TRIAL: NCT00822250
Title: Clinical and Biological Study of Sub-pigmentation During Infantile Cystinosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Département de la Recherche Clinique et de l'Innovation, CHU de Nice
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 07-PP-05
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-10

CONDITIONS: Cystinosis
MeSH Terms: conditions — Cystinosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): cutting hair, skin phenotype description
  Interventions: Other: analysis of pigmentation

INTERVENTIONS:
Other: analysis of pigmentation — cutting hair, skin description, skin biopsy for only 4 patients
  Other Names: surgical biopsy; skin examination

SUMMARY:
The purpose of this study is to determine the molecular mechanism of this disease and to research the relationship between cystinosis and skin phenotype.

ELIGIBILITY:
Inclusion Criteria:

1. cystinosis
2. known CTNS mutation

Exclusion Criteria:

1. patient with corticotherapy treatment
2. patient with immunosuppressant treatment

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
to determine molecular mechanism of the disease | at time= 0

SECONDARY OUTCOMES:
to research relationship between skin phenotype and cystinosis | at time =0

CONTACTS AND LOCATIONS:
Locations (1):
- department of dermatology, Nice University Hospital, Nice, France